CLINICAL TRIAL: NCT00667420
Title: A Pilot Study of Perioperative Panitumumab in Combination With Epirubicin, Oxaliplatin and Xeloda in Patients With Resectable Gastroesophageal Adenocarcinoma
Brief Title: Perioperative Panitumumab and Epirubicin, Oxaliplatin and Xeloda (EOX) in Patients With Gastroesophageal Adenocarcinoma
Acronym: EOXP
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Closed due to slow accrual
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David Patrick Ryan, MD, Clinical Director, MGH Cancer Center, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07326
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Esophageal Adenocarcinoma; Gastric Adenocarcinoma
Keywords: gastric; esophageal; panitumumab
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — Panitumumab; Epirubicin; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EOXP chemotherapy (Experimental): open-label, single-arm EOXP Epirubicin 50mg/m2 by IV on day 1 of each 21 day cycle, Oxaliplatin 100 mg/m2 by IV on day 1 of each 21 day cycle, Capecitabine 400 mg/m2 twice daily by mouth on days 1-21 of the 21 day cycle Panitumumab - 9mg/kg by IV on day 1 of each 21 day cycle
  Interventions: Drug: panitumumab, epirubicin, oxaliplatin, xeloda

INTERVENTIONS:
Drug: panitumumab, epirubicin, oxaliplatin, xeloda — pilot study

SUMMARY:
A pilot study to determine the safety of using perioperative panitumumab with EOX (epirubicin, oxaliplatin, and capecitabine) in patients with adenocarcinoma of the esophagus and stomach.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of adenocarcinoma of the stomach, gastroesophageal junction, or lower third of the esophagus, AJCC stage II-IIIB (gastric) or IIA-IVA (esophageal). M1a disease will be included, but not T4 lesions.
* No prior radiation or chemotherapy including anti-EGFR or vascular endothelial growth factor (VEGF) antibody or tyrosine kinase inhibitor treatments.
* All patients must have staging endoscopic ultrasound (EUS) prior to enrollment.
* Men or Women >18 years of Age
* ECOG performance status <2 (Karnofsky >60%, see Appendix A).
* Cardiac ejection fraction >45% by echocardiogram or MUGA scan.
* Must be able to either swallow pills or have gastrostomy tube in place for administration of enteral medications.
* Patients must have normal organ, metabolic and marrow function as defined below:

  * Hematologic function, as follows:

    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * Platelet count ≥ 100 x 109/L
    * Hemoglobin ≥ 9.0 g/dL
  * Renal function, as follows:

    * Creatinine < or = 1.5 mg/dL x ULN

Hepatic function, as follows:

* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT)< or = 3 x ULN
* Total bilirubin < 1.5 x ULN

Metabolic function, as follows:

* Magnesium ≥ lower limit of normal
* Calcium < or = lower limit of normal -Human IgG is known to cross the placental barrier; therefore, Panitumumab may be transmitted from the mother to the developing fetus. In women of childbearing potential, appropriate contraceptive measures must be used during treatment with panitumumab and for 6 months following the last dose of panitumumab. If panitumumab is used during pregnancy or if the patient becomes pregnant while receiving this drug, she should be apprised of the potential risk for loss of the pregnancy or potential hazard to the fetus.

3.1.10 Ability to understand and the willingness to sign and date a written IEC/IRB approved informed consent form.

Exclusion Criteria:

* Evidence of distant metastatic disease.
* T4 tumor on initial staging studies.
* History of another primary cancer, except:
* Curatively treated in situ cervical cancer
* Curatively resected non-melanoma skin cancer
* Other primary solid tumor curatively treated with no known active disease present and no treatment administered for ³ 5 years prior to enrollment
* Relative or absolute contraindications to surgery which in the opinion of the investigator make the patient a poor candidate for surgical resection.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to panitumumab or other agents used in study.
* Subjects requiring chronic use of immunosuppressive agents (e.g., methotrexate, cyclosporine).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or any evidence of interstitial lung disease on baseline chest CT scan.
* History of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risks associated with the study participation or investigational product(s) administration or may interfere with the interpretation of the results.
* Subject unwilling or unable to comply with study requirements.
* Women who test positive for serum or urine pregnancy test < 72 hours before randomization or are breast feeding.
* Known positive test(s) for human immunodeficiency virus infection, hepatitis C virus, acute or chronic active hepatitis B infection.
* Major surgery with 28 days or minor surgery within 14 days of study enrollment.
* Men or women of child-bearing potential (women who are post-menopausal < 52 weeks, not surgically sterilized, or not abstinent) not consenting to use adequate contraception (per institutional standard of care) during the course of the study and after the last investigational product(s) administration (24 weeks for women, 4 weeks for men).
* Subjects with > grade 1 neuropathy at baseline.
* Contraindication to port-a-cath placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-04; Primary Completion 2011-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Ryan, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - DFCI, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 2008 and July 2010, 17 patients with adenocarcinoma of the stomach were accrued to the protocol at the MGH and Dana Farber Cancer Institute.
Groups:
- Epirubicin, Oxaliplatin, Capecitabine, Panitumumab Treatment: Panitumumab in Combination with Epirubicin, Oxaliplatin and Capecitabine (EOX-P)
Period: Overall Study
Arm/Group | Epirubicin, Oxaliplatin, Capecitabine, Panitumumab Treatment
Started | 17
Completion of Pre-operative EOX-P | 15
Completion of Surgery/Re-staging | 11
Completed | 7
Not Completed | 10
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 5
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 17 patients with adenocarcinoma of the stomach were enrolled on this study of perioperative EOX-P.
Arm/Group | Epirubicin, Oxaliplatin, Capecitabine, Panitumumab Treatment
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 59 (NA) [40 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Safety and tolerability were measured by assessing the number of participants able to complete 3 cycles of pre-operative chemotherapy
Time Frame: after 3 cycles of pre-operative chemotherapy (approx 21 days per cycle)
Measure: Number; unit: participants
Arm/Group | Epirubicin, Oxaliplatin, Capecitabine, Panitumumab Treatment
Number analyzed (Participants) | 17
participants | 14

2. Secondary Outcome: R0 Resection Rate
Description: percentage of participants who have microscopically negative margins (no tumor at/near the edge of what is resected) at the time of surgical resection
Time Frame: time of surgery = after 3 cycles (approx 63 days) of pre-operative EOX-P chemotherapy
Measure: Number; unit: percentage of participants
Groups:
- Epirubicin, Oxaliplatin, Capecitabine, Panitumumab Treatment: Panitumumab in Combination with Epirubicin, Oxaliplatin, and Capecitabine (EOX-P) Chemotherapy.
Arm/Group | Epirubicin, Oxaliplatin, Capecitabine, Panitumumab Treatment
Number analyzed (Participants) | 17
percentage of participants | 52.9 [lower limit 1]

3. Secondary Outcome: Progression-Free Survival
Description: measured from the first day of treatment to the day when conclusive evidence of new disease is found
Time Frame: up to 72 months
Population: We enrolled 17 patients
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Epirubicin, Oxaliplatin, Capecitabine, Panitumumab Treatment
Number analyzed (Participants) | 17
months | 27.2 (24.2)

4. Secondary Outcome: Pathologic Complete Response Rate
Description: For patients who undergo complete resection, those who have no evidence of residual viable tumor in the surgical specimen will be declared to have achieved a complete pathologic response (pCR), and the overall percentage of patients with pCR will be determined.
Time Frame: at surgical resection, after 3 cycles pre-operative chemotherapy (approx 63 days)
Measure: Number; unit: participants
Arm/Group | Epirubicin, Oxaliplatin, Capecitabine, Panitumumab Treatment
Number analyzed (Participants) | 12
participants | 0

5. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is the duration from start of treatment to time of death from any cause.
Time Frame: duration from enrollment to death (up to 6 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Epirubicin, Oxaliplatin, Capecitabine, Panitumumab Treatment
Number analyzed (Participants) | 17
months | NA [NA to NA] — At time study was closed, this regimen was not to be used in this patient population and therefore overall survival was not followed.

ADVERSE EVENTS:
Time Frame: From start of study drug (day 1) throughout time enrolled on study. (June 2008 - January 2011)
Description: Adverse events seen in this study were not significantly different from those reported by Waddell T, et. al in Lancet Oncol. 2013 May;14(6):481-9. (NCT00824785). Therefore, only grade 3 and 4 adverse events have been reported here.
Arm/Group | Epirubicin, Oxaliplatin, Capecitabine, Panitumumab Treatment
Serious Adverse Events (participants affected / at risk) | 6/17
Other Adverse Events (participants affected / at risk) | 13/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epirubicin, Oxaliplatin, Capecitabine, Panitumumab Treatment (N=17)
Amylase (Metabolism and nutrition disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Infection - bacteremia (Infections and infestations) | 1
Lipase (Metabolism and nutrition disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Tachycardia (Cardiac disorders) | 1
diarrhea (Gastrointestinal disorders) | 2
hypocalcemia (Metabolism and nutrition disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epirubicin, Oxaliplatin, Capecitabine, Panitumumab Treatment (N=17)
Elevated SGPT (Metabolism and nutrition disorders) | 1 (3)
Elevated SGOT (Metabolism and nutrition disorders) | 2 (3)
Abdomen - pain (Gastrointestinal disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 3 (4)
Dehydration (Gastrointestinal disorders) | 3 (4)
Diarrhea without prior colostomy (Gastrointestinal disorders) | 3 (4)
Febrile neutropenia (Infections and infestations) | 2 (2)
Fistula - esophageal (Gastrointestinal disorders) | 1 (1)
Hemoglobin - low (Blood and lymphatic system disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 6 (7)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (7)
Hypotension (Cardiac disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection - lung (Infections and infestations) | 1 (1)
Leak - incl. anastomotic - esophagus (Gastrointestinal disorders) | 1 (1)
Leukocytes - low (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Neutrophils (Blood and lymphatic system disorders) | 3 (4)
Platelets - low (Blood and lymphatic system disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 1 (1)
Weight loss (General disorders) | 2 (4)

LIMITATIONS AND CAVEATS:
This study was stopped early due to poor tolerability. We will not further study this regimen in this patient population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No